CLINICAL TRIAL: NCT01308723
Title: Exploratory Open Label Dose-escalation Phase Ib Study to Evaluate Safety, Pharmacokinetics and Therapeutic Activity of RO5323441, Administered Intravenously, in Combination With Sorafenib (Nexavar®), in Patients With Advanced or Metastatic and/or Unresectable Hepatocellular Carcinoma
Brief Title: A Dose-Finding and Exploratory Study of RO5323441 in Combination With Sorafenib in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP25497
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — TB-403; Sorafenib

ARMS (3):
- Part I (Experimental)
  Interventions: Drug: RO5323441; Drug: sorafenib
- Part II (A) (Experimental)
  Interventions: Drug: RO5323441; Drug: sorafenib
- Part II (B) (Active Comparator)
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: RO5323441 — escalating doses iv
  Arms: Part I
Drug: RO5323441 — iv every 2 weeks
  Arms: Part II (A)
Drug: sorafenib — 400 mg orally twice daily to once every other day

SUMMARY:
This open-label study will assess the safety, efficacy and pharmacokinetics of RO5323441 in combination with sorafenib in patients with advanced or metastatic hepatocellular carcinoma previously untreated with systemic therapy. In the dose-finding Part I, cohorts of patients will receive escalating doses of RO5323441 intravenously (iv) every 2 weeks in combination with sorafenib 400 mg orally twice daily. In the exploratory Part II, patients will be randomized to receive either the previously established dose of RO5323441 iv every 2 weeks plus continuous oral sorafenib or sorafenib alone. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs. For patients in the sorafenib arm with disease progression crossover to combination treatment with RO5323441 will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 21 years of age
* Advanced or metastatic and/or unresectable hepatocellular carcinoma
* At least 1 measurable lesion according to RECIST criteria
* Primary tumor in situ (Expansion Cohort Part I, Part II)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Prior systemic treatment for metastatic hepatocellular carcinoma or patients who had tumor removed (Expansion Cohort Part I, Part II)
* Major surgery within previous 4 weeks or planned major surgical procedure during course of study
* Radiation therapy within 28 days prior to start of study treatment
* Serious non-healing wound, ulcer ore bone fracture
* History of uncontrolled seizures or encephalopathy within the last 6 months
* Current central nervous system (CNS) metastases or spinal cord compression
* History of gastrointestinal perforation or esophageal/gastric bleeding within 6 months prior to study enrollment
* History of another primary malignancy and off treatment for </= 3 years, except for non-melanoma skin cancer and carcinoma in situ of the cervix
* Patients with prior liver transplant
* Inadequately controlled hypertension or prior history of hypertensive crisis or hypertensive encephalopathy
* Active bleeding diathesis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Part I : Safety/dose-limiting toxicity: Incidence of adverse events | up to 12 months
Part I: Determination of recommended Part II dose | up to 12 months
Part II: Safety/tolerability: Incidence of adverse events | up to 28 months

SECONDARY OUTCOMES:
Pharmacokinetics of RO5323441 in combination with sorafenib | up to 40 months
Pharmacokinetics of sorafenib in combination with RO5323441 | up to 12 months
Pharmacodynamic biomarkers (DCE-Magnetic Resonance Imaging evaluations, Placental Growth Factor, Vascular Endothelial Growth Factor Receptors) | up to 40 months
Efficacy: tumor assessments by Magnetic Resonance Imaging or Computed Tomography according to RECIST criteria | up to 40 months
Impact on wound healing (skin biopsies) | up to 40 months
Safety: additional anti-drug antibodies sampling after termination of study drug treatment | 2 and 4 months after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Singapore, Singapore